CLINICAL TRIAL: NCT03856684
Title: Randomized Trial Evaluating Women's Behavior Not Participating in Cervical Cancer Screening Facing Three Strategies for Optimizing Home Sending by Post of Vaginal Self-sampling Kit
Brief Title: Evaluation of Three Strategies Based on Vaginal Self-sampling Kit Send to Home of Unscreened Women for Cervical Cancer
Acronym: APACHE-4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Centre Régional de Coordination des Dépistages des Cancers - Centre-Val de Loire (Unknown); Centre d'Investigation Clinique-P1415, TOURS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DR170135-APACHE-4
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Cervical Cancer Screening; Cervical Cancer
Keywords: vaginal; self-sampling; cervical cancer screening; Papillomavirus; HPV; High Risk Human papillomavirus Infection; pap smear
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self-sampling kit sent at home (Active Comparator): Sending of a vaginal self-sampling kit at home
  Interventions: Behavioral: Self-sampling kit sent at home
- Self-sampling kit sent at home + SMS reminder (Experimental): Sending of a vaginal self-sampling kit at home + a SMS reminder is sent if the woman do not (in 2 months) :
  * perform a pap smear
  * or send her vaginal self-sample to the laboratory
  * or contact the screening center to inform to an exclusion reason
  Interventions: Behavioral: Self-sampling kit sent at home + SMS reminder
- Letter offering a self-sampling kit "on request"+ SMS reminder (Experimental): Sending of letter offering a vaginal self-sampling kit. Women can ask for this kit on line, on our website or by calling us.
  If they do ask for the kit, one kit is sending to their home.
  For these women, a SMS reminder is sent if the woman do not (in 2 months) :
  * perform a pap smear
  * or send her vaginal self-sample to the laboratory
  * or contact the screening center to inform to an exclusion reason
  Interventions: Behavioral: Letter offering a self-sampling kit "on request"+ SMS reminder
- SMS offering a self-sampling kit "on request"+ SMS reminder (Experimental): Sending of SMS offering a vaginal self-sampling kit. Women can ask for this kit on line, on our website or by calling us.
  If they do ask for the kit, one kit is sending to their home.
  For these women, a SMS reminder is sent if the woman do not (in 2 months) :
  * perform a pap smear
  * or send her vaginal self-sample to the laboratory
  * or contact the screening center to inform to an exclusion reason
  Interventions: Behavioral: SMS offering a self-sampling kit "on request"+ SMS reminder

INTERVENTIONS:
Behavioral: Self-sampling kit sent at home — Selected women receive a mail inviting them either to perform a vaginal self sampling at their home (with the kit provided) or to perform a pap smear.
  When women choose the vaginal self-sampling, a HPV test is performed on the sample in a virology laboratory.
  Arms: Self-sampling kit sent at home
Behavioral: Self-sampling kit sent at home + SMS reminder — Selected women receive a mail inviting them either to perform a vaginal self sampling at their home (with the kit provided) or to perform a pap smear.
  After 2 months without "return", a SMS reminder about the available self-sampling kit is sent to the woman. We call "return" :
  * the receipt of the vaginal self-sample at the laboratory
  * the performance of a pap smear
  * Information about recent screening test or a cervical screening exclusion reason When women choose the vaginal self-sampling, a HPV test is performed on the sample in a virology laboratory.
  Arms: Self-sampling kit sent at home + SMS reminder
Behavioral: Letter offering a self-sampling kit "on request"+ SMS reminder — Selected women receive a mail inviting them either to perform a vaginal self sampling at their home (kit provided on request) or to perform a pap smear.
  Women are invited to ask the kit online, on our website.
  For the women who ask the kit, after 2 months without "return", a SMS reminder about the available self-sampling kit is sent to the woman. We call "return" :
  * the receipt of the vaginal self-sample at the laboratory
  * the performance of a pap smear
  * Information about recent screening test or a cervical screening exclusion reason When women choose the vaginal self-sampling, a HPV test is performed on the sample in a virology laboratory.
  Arms: Letter offering a self-sampling kit "on request"+ SMS reminder
Behavioral: SMS offering a self-sampling kit "on request"+ SMS reminder — Selected women receive a SMS inviting them to ask a vaginal self sampling kit to perform a sample at home and send it to a laboratory (kit provided on request).
  Women are invited to ask the kit by answering "1" by SMS.
  For the women who ask the kit, after 2 months without "return", a SMS reminder about the available self-sampling kit is sent to the woman. We call "return" :
  * the receipt of the vaginal self-sample at the laboratory
  * the performance of a pap smear
  * Information about recent screening test or a cervical screening exclusion reason When women choose the vaginal self-sampling, a HPV test is performed on the sample in a virology laboratory.
  Arms: SMS offering a self-sampling kit "on request"+ SMS reminder

SUMMARY:
Despite the existence of an effective screening test (pap smear), cervical cancer is, every year in France, the cause of more than 3,000 new cases and 1,100 deaths. But, in France, 4 in 10 women are not screened or not often enough (nearly 7 millions women). It is therefore necessary to develop new strategies to reach these women. The etiological factor of this cancer is persistent infection with High-Risk Human PapillomaVirus (HR-HPV). Thereby, HPV-based tests could be alternative screening tests. Vaginal self-sampling with HR-HPV test is simpler and less intrusive than the pap smear. It has been shown that sending vaginal self-sampling kit (with HPV test) to unscreened women's home is a powerful means to increase the participation rate of cervical cancer screening. It seems interesting to explore methods to increase the efficiency of this strategy by optimizing the ratio of the number of kits used compared to the number of kits sent. Two approaches will be tested: a system "available on request" of the kit and / or the addition of an SMS (Short Message Service) reminder.

ELIGIBILITY:
Inclusion Criteria:

* women from 30 to 66 years old
* women living in french territorial division 37 ("Indre-et-Loire")
* women with a mobile phone in database
* women who do not perform a pap smear in the last 4 years
* women who do not answer to a first "invitation" letter to perform a pap smear

Exclusion Criteria:

* STOP SMS
* HPV cervical pathology during treatment
* Hysterectomy including cervix

Ages: 30 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10400 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Participation / no participation to complete cervical cancer screening | 9 months after postal mail (with or without the kit) or SMS
  Complete cervical cancer screening is defined as one of the followings :
  * perform a pap smear
  * perform a vaginal self-sampling with negative HR-HPV test
  * perform a vaginal self-sampling with noninterpretable HR-HPV test result followed by a control pap smear (nine-month extension to do the pap smear after the sending of the HPV result)
  * perform a vaginal self-sampling with positive HR-HPV test result followed by a control pap smear (nine-month extension to do the pap smear after the sending of the HPV result)

CONTACTS AND LOCATIONS:
Overall Officials: Julie BOYARD, MSc, Principal Investigator — University Hospital of TOURS
Locations (1):
- Crcdc-Cvl, Tours, France

IPD SHARING:
Plan to Share IPD: No